CLINICAL TRIAL: NCT02291523
Title: The Effect of Therapeutic Fecal Transplant on the Gut Microbiome in Children With Ulcerative Colitis
Acronym: FMT_UC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Sonia Michail, MD, Professor of Clinical Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHLA-16-00050
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Ulcerative Colitis
Keywords: Fecal transplant
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patient Stool Transplant (Sham Comparator): Arm 1 will get FMT (Fecal Microbial Transplant) placebo and high dose 5-ASA (Pentasa). The FMT is done through colonoscopy.
  Interventions: Biological: Fecal Microbial Transplant
- Donor Stool Transplant (Active Comparator): Arm 2 will get FMT (Fecal Microbial Transplant) with Healthy Donor Stool and high dose 5-ASA (Pentasa). The FMT is done through colonoscopy.
  Interventions: Biological: Fecal Microbial Transplant

INTERVENTIONS:
Biological: Fecal Microbial Transplant — Fecal Transplant via Colonoscopy.
  Other Names: FMT

SUMMARY:
Ninety Six patients with mild to moderate ulcerative colitis will be randomized to double blind, placebo controlled study. The safety and efficacy of the intervention will be closely monitored.

DETAILED DESCRIPTION:
The enteric microbiota is now accepted as an important etiologic factor in the pathogenesis of human Inflammatory Bowel Disease (IBD) and immune-mediated chronic experimental intestinal inflammation, with ample data to implicate the microbiome as a main factor in the occurrence of IBD. This can be inferred from animals in germ-free environment which can protect from experimental colitis. In addition, increased gut permeability due to dysbiosis, is frequently seen in patients with IBD even in remission and, similarly, first degree relatives of IBD. Therefore, it is not surprising that therapeutic interventions aiming at modifying the gut microbiome would be of therapeutic benefit. Ulcerative colitis is a condition that is characterized by chronic inflammation of the colon. It is an important pediatric disease as 25% of all cases begin in childhood and its incidence is continuously on the rise. It is believed to be related to a genetically and environmentally-generated altered immune response to the enteric microbiome. Previous work in the PI's laboratory suggests that children harbor a unique gut microbial profile, which can predict therapeutic response. Therefore, modifying the gut microbiome may result in therapeutic benefit. However, attempts to modify the gut microbiome were largely unsuccessful until the advent of fecal transplant, which is a new approach in treating colitis. Fecal microbiota transplant (FMT) has been introduced several decades ago in an attempt to restore the gut microbial balance and it appears to be a more efficient method to effectively change and sustain the gut microbial composition. To date there have been a number of successful reports to suggest control of disease activity and in some cases cure of the disease. This study aims to further determine the safety and efficacy of FMT in treating children with ulcerative colitis

ELIGIBILITY:
Inclusion Criteria

* Age: 7-21 who have been diagnosed with ulcerative colitis
* Mild to moderate disease based on PUCAI with a score of 10-64
* Need for colonoscopy

Exclusion Criteria

* Children who are known to be resistant to steroid therapy, immunomodulators and biologics, or on a steroid dose greater than 0.5 mg/kg/day (maximum 20 mg)
* Children with recent dose change of biologics (within 4 weeks), 5-ASA, steroids or immunomodulators (within 4 weeks)
* Allergy to or intolerance of mesalamine or 5-ASA products
* Any evidence of infectious colitis
* Concurrent infections that require anti-microbial therapy (such as abdominal abscess, pneumonia, etc…)
* Unable to give informed consent/assent
* Have received probiotic preparations ≤ 4 weeks prior to randomization
* Pregnancy and breast feeding in patient subjects of childbearing potential
* Subjects with significant renal and liver dysfunction (creatinine > 2 mg/dl and direct bilirubin > 2 mg/dl), Subjects with congenital or acquired immunodeficiency, or who are immunosuppressed due to conditions other than ulcerative colitis (such as neoplastic disease or organ transplantation), have received or are receiving chemotherapy, or have been diagnosed with HIV.

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 101 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is disease remission based on PUCAI scores (<10). | 12 Months
  The primary outcome including results of disease activity, and safety measures.

SECONDARY OUTCOMES:
Secondary endpoints will include change in mucosal inflammation reflected on laboratory studies. | 12 Months
  Secondary endpoints include changes in gut microbial diversity - determined by gut microbial genomics and proteomics, and outcome measures for mucosal inflammation and repair including laboratory testing such as the level for C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR) as well as the stool calprotectin level.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Michail, MD, Principal Investigator — Children Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michail S, Bultron G, Depaolo RW. Genetic variants associated with Crohn's disease. Appl Clin Genet. 2013 Jul 16;6:25-32. doi: 10.2147/TACG.S33966. Print 2013. PMID 23935379
- [Background] Michail S, Durbin M, Turner D, Griffiths AM, Mack DR, Hyams J, Leleiko N, Kenche H, Stolfi A, Wine E. Alterations in the gut microbiome of children with severe ulcerative colitis. Inflamm Bowel Dis. 2012 Oct;18(10):1799-808. doi: 10.1002/ibd.22860. Epub 2011 Dec 14. PMID 22170749
- [Background] Hyams JS, Lerer T, Mack D, Bousvaros A, Griffiths A, Rosh J, Otley A, Evans J, Stephens M, Kay M, Keljo D, Pfefferkorn M, Saeed S, Crandall W, Michail S, Kappelman MD, Grossman A, Samson C, Sudel B, Oliva-Hemker M, Leleiko N, Markowitz J; Pediatric Infl ammatory Bowel Disease Collaborative Research Group Registry. Outcome following thiopurine use in children with ulcerative colitis: a prospective multicenter registry study. Am J Gastroenterol. 2011 May;106(5):981-7. doi: 10.1038/ajg.2010.493. Epub 2011 Jan 11. PMID 21224840
- [Derived] Le J, Hakimjavadi H, Parsana R, Chamala S, Michail S. Fecal Microbiota Transplantation Induces Sustained Gut Microbiome Changes in Pediatric Ulcerative Colitis: A Combined Randomized and Open-Label Study. Gastro Hep Adv. 2025 Jul 11;4(10):100741. doi: 10.1016/j.gastha.2025.100741. eCollection 2025. PMID 40933007